CLINICAL TRIAL: NCT05891470
Title: A Randomized Phase II Study to Explore the Benefits of the MonaLisa Touch® System in the Improvement of the Sexual QUAlity of Life in Gynaecological Cancer Patients Treated by (Chemo)-Radiotherapy.(SQUAL)
Brief Title: To Explore the Benefits of the MonaLisa Touch® System in Gynaecological Cancer Patients Treated by (Chemo)-RT
Acronym: SQUAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Principal Investigator, Clémence Al Wardi, Pr, Jules Bordet Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE3596
Record Dates: First submitted 2023-04-17; First posted 2023-06-07 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Gynecologic Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Vaginal Dilatators (Active Comparator): Use of vaginal dilatators as standard of care.
  Interventions: Device: Vaginal dilatators
- MonaLisa Touch device (Experimental): Sessions with the MonaLisa Touch device
  Interventions: Device: MonaLisa Touch device

INTERVENTIONS:
Device: MonaLisa Touch device — sessions with intra-vaginal CO2 laster system
  Arms: MonaLisa Touch device
Device: Vaginal dilatators — Home use of vaginal dilatators (at least twice a week for minimum 5 minutes)
  Arms: Vaginal Dilatators

SUMMARY:
The increasing survival rate of gynaecological cancer patients highlights the need to improve their Quality of Life (QoL) after treatment. Among all QoL factors, sexuality is unfortunately often neglected, especially vaginal dryness and fibrosis/stenosis. Currently, the latter is standardly treated by vaginal dilators, which may induce pain and discomfort (1). A new possibility, already used in some centers, is the MonaLisa Touch® system, a microablative CO2 laser (2). Its efficiency to improve sexual QoL has already been demonstrated in breast cancer patients treated with chemotherapy and/or hormonotherapy and in menopausal women (3). Unfortunately, almost no study have been conducted yet for patients undergoing radiotherapy to the pelvic area to prevent vaginal morbidity. Our randomised study will explore the benefits of the MonaLisa Touch® device for the prevention of sexual adverse events induced by pelvic (chemo-) radiotherapy for pelvic cancers.

DETAILED DESCRIPTION:
Patients will be randomly (1:1) assigned to the dilators (standard of care) or MonaLisa Touch® system (2 arms). Patients will be stratified for endometrial or cervix cancer, radiotherapy dose and techniques, menopausal status, tumor stage, chemotherapy or not, surgery or not. Patients will begin the Mona Lisa at 3 months, once per month during 6 months while the follow-up assessment will continue until 12M after end of RT treatment. Patients randomized in dilator arm will also begin 3 months post end of RT and will use them twice every 2 weeks for 12M (as standard of care).

Questionnaires (FSFI- Female Sexual Function Index [10], SHQ-22) and VHI (Vaginal Health Index [11]) will be performed before treatment, at 3, 6, 9, 12 and 15M. Partners will also be asked to fill the sexual quality of life questionnaire EORTC SHQ-22 before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* (chemo)radiotherapy +/- brachytherapy, gynaecologic cancer patients
* complete response on the imagery at 3 months (PET scan/MRI).
* Stades I-III

Exclusion Criteria:

* M1
* Stade IV
* No complete response under imagery at 3months
* Relapse of gynaecological cancer
* Active gynaecological infection
* Pelvic organ prolapse more than stage II
* Local vaginal hormone therapy within 6 weeks prior to enrolment

Max Age: 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-02-02 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Variations of the sexual function through FSFI questionnaire | before (chemo-RT) to 15 months post (Chemo)-RT treatment
  Sexual QOL questionnaire
Variations of the sexual function through SHQ-22 questionnaire | before (chemo-RT) to 15 months post (Chemo)-RT treatment
  Sexual QOL questionnaire

SECONDARY OUTCOMES:
Vaginal functional changes by means of VHI score | 3 months to 15 months post (Chemo)-RT treatment
  Objective assessement through vaginal tactus
Patient complience | 3 months to 15 months post (Chemo)-RT treatment
  Percentage of patients who followed the required treatment as required.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Van Gestel, Pr, MD, PhD, Study Director — Jules Bordet Institute
Locations (1):
- Institut Jules Bordet, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No